CLINICAL TRIAL: NCT00428454
Title: A Randomized Comparison of Sirolimus-eluting Stent Implantation With Zotarolimus-eluting Stent Implantation for the Treatment of Chronic Total Coronary Occlusions. The PRISON III Trial.
Brief Title: Sirolimus-eluting vs Zotarolimus-eluting Stents for Chronic Total Coronary Occlusions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R&D Cardiologie (Other)
Collaborators: Cordis US Corp. (Industry)
Responsible Party: Principal Investigator, Dr. M.J. Suttorp, MD, PhD, FESC, FACC, R&D Cardiologie
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDC-2006-02
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Coronary Artery Disease; Coronary Disease; Coronary Stenosis
Keywords: drug-eluting stent; chronic total occlusion; sirolimus-eluting stent; zotarolimus-eluting stent; QCA
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Zotarolimus eluting stent (Experimental): Zotarolimus eluting stent
  Interventions: Device: sirolimus-eluting stent, zotarolimus-eluting stent
- Sirolimus eluting stent (Active Comparator): Sirolimus eluting stent
  Interventions: Device: sirolimus-eluting stent, zotarolimus-eluting stent

INTERVENTIONS:
Device: sirolimus-eluting stent, zotarolimus-eluting stent — PCI in chronically occluded coronary artery

SUMMARY:
Primary intracoronary stent placement after successfully crossing chronic total coronary occlusions (CTO) decreases the high restenosis rate at long-term follow-up compared with conventional balloon angioplasty. Several studies have shown the efficacy of sirolimus-eluting stents in selected groups of patients. In the PRISON II study we demonstrated that sirolimus-eluting stents were superior to bare metal stents in CTO. In this prospective randomized trial, sirolimus-stent implantation will be compared with zotarolimus-eluting stent implantation for the treatment of chronic total coronary occlusions. A total of 300 patients will be clinically followed up for 1, 6, 12 months, 2, 3, 4, 5 year with angiographic follow-up at 8 months. Quantitative coronary analysis will be performed by an independent core laboratory. The primary end point is in-segment late luminal loss at 8 month angiographic follow-up.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) of chronic total occlusions (CTO) was traditionally limited by high restenosis rates. Coronary stenting using bare metal stents significantly decreases restenosis in CTO compared to balloon angioplasty alone, but restenosis rates still reach 32-55%. In 200 patients with CTO, randomized in the PRISON I study we demonstrated a restenosis rate of 22% after bare metal stent (BMS) implantation as compared with 33% after conventional balloon angioplasty. During the past few years, sirolimus (rapamycin), a cytostatic macrocyclic lactone with anti-inflammatory and antiproliferative properties, delivered from a polymer-encapsulated stent was shown to almost eliminate the risk of restenosis in selected groups of patients. The drug zotarolimus (ABT-578), a sirolimus analogue, is designed to inhibit the cellular process that leads to restenosis. In the PRISON II study we have randomized 200 patients with CTO to either BMS implantation or sirolimus-eluting stent implantation and we demonstrated a reduction of in-stent binary restenosis from 36% to 7% and in-segment binary restenosis rates from 41% to 11% in favour of the sirolimus eluting stent. However, no data are available on direct comparison of the clinical efficacy, safety, and angiographic outcome of particular drug-eluting stents in patients with CTO and there may be differences between various drug-eluting stents. The PRISON III study is designed to address this issue and provide information about two different drug-eluting stents. It is a prospective randomized, single blinded trial comparing the relative safety, clinical efficacy and angiographic outcomes of sirolimus and zotarolimus-eluting stents in patients undergoing successful recanalization of CTO.

ELIGIBILITY:
INCLUSION CRITERIA

* the estimated duration of the occlusion is at least 2 weeks.
* signs of ischemia related to the occluded coronary artery.
* successful recanalization of the occluded artery is achieved.
* reference diameter is > 2.5 mm.
* written informed consent obtained.

EXCLUSION CRITERIA

* primary or rescue PCI for acute myocardial infarction
* the lesion could not be crossed.
* lesions with complex anatomy making successful stent deployment unlikely.
* the guide wire is not in the true lumen distal to the occlusion.
* Sirolimus or zotarolimus allergy
* venous or arterial bypass grafts
* pregnant or nursing women.
* participation in an other trial.
* factors making long-term follow-up difficult or unlikely.
* life expectancy <1 year.
* contraindications for ASA or Clopidogrel or heparin.
* use of coumadins that could not be stopped before the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
In-segment late luminal loss at 8 months as assessed by an independent angiographic core lab. | 8 month

SECONDARY OUTCOMES:
In-stent late luminal loss | 8 month
In-stent and in-segment binary restenosis rate | 8 month
In-stent and in-segment MLD | 8 month
Percentage diameter stenosis | 8 month
A composite of major adverse cardiac events (MACE: death, myocardial infarction and clinically driven target lesion revascularization) | 8 month
Stent thrombosis (acute, <1day; subacute, 1 to 30 days; and late, >30 days) | 30 days
Target vessel failure up to 5 year of clinical follow-up. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Maarten J. Suttorp, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (5):
- AZ Middelheim, Antwerp, Antwerpen, Belgium
- Netherlands (4):
  - AMC, Amsterdam, Amsterdam
  - Catharina Ziekenhuis, Eindhoven, Eindhoven
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - St Antonius Hospital, Nieuwegein

REFERENCES:
- [Background] Rahel BM, Suttorp MJ, Laarman GJ, Kiemeneij F, Bal ET, Rensing BJ, Ernst SM, ten Berg JM, Kelder JC, Plokker HW. Primary stenting of occluded native coronary arteries: final results of the Primary Stenting of Occluded Native Coronary Arteries (PRISON) study. Am Heart J. 2004 May;147(5):e22. doi: 10.1016/j.ahj.2003.11.023. PMID 15131557
- [Background] Suttorp MJ, Mast EG, Plokker HW, Kelder JC, Ernst SM, Bal ET. Primary coronary stenting after successful balloon angioplasty of chronic total occlusions: a single-center experience. Am Heart J. 1998 Feb;135(2 Pt 1):318-22. doi: 10.1016/s0002-8703(98)70099-7. PMID 9489982
- [Background] Serruys PW, de Jaegere P, Kiemeneij F, Macaya C, Rutsch W, Heyndrickx G, Emanuelsson H, Marco J, Legrand V, Materne P, et al. A comparison of balloon-expandable-stent implantation with balloon angioplasty in patients with coronary artery disease. Benestent Study Group. N Engl J Med. 1994 Aug 25;331(8):489-95. doi: 10.1056/NEJM199408253310801. PMID 8041413
- [Background] Fischman DL, Leon MB, Baim DS, Schatz RA, Savage MP, Penn I, Detre K, Veltri L, Ricci D, Nobuyoshi M, et al. A randomized comparison of coronary-stent placement and balloon angioplasty in the treatment of coronary artery disease. Stent Restenosis Study Investigators. N Engl J Med. 1994 Aug 25;331(8):496-501. doi: 10.1056/NEJM199408253310802. PMID 8041414
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Sirnes PA, Golf S, Myreng Y, Molstad P, Emanuelsson H, Albertsson P, Brekke M, Mangschau A, Endresen K, Kjekshus J. Stenting in Chronic Coronary Occlusion (SICCO): a randomized, controlled trial of adding stent implantation after successful angioplasty. J Am Coll Cardiol. 1996 Nov 15;28(6):1444-51. doi: 10.1016/s0735-1097(96)00349-x. PMID 8917256
- [Background] Suttorp MJ, Laarman GJ, Rahel BM, Kelder JC, Bosschaert MA, Kiemeneij F, Ten Berg JM, Bal ET, Rensing BJ, Eefting FD, Mast EG. Primary Stenting of Totally Occluded Native Coronary Arteries II (PRISON II): a randomized comparison of bare metal stent implantation with sirolimus-eluting stent implantation for the treatment of total coronary occlusions. Circulation. 2006 Aug 29;114(9):921-8. doi: 10.1161/CIRCULATIONAHA.106.613588. Epub 2006 Aug 14. PMID 16908768
- [Background] Kandzari DE, Leon MB, Popma JJ, Fitzgerald PJ, O'Shaughnessy C, Ball MW, Turco M, Applegate RJ, Gurbel PA, Midei MG, Badre SS, Mauri L, Thompson KP, LeNarz LA, Kuntz RE; ENDEAVOR III Investigators. Comparison of zotarolimus-eluting and sirolimus-eluting stents in patients with native coronary artery disease: a randomized controlled trial. J Am Coll Cardiol. 2006 Dec 19;48(12):2440-7. doi: 10.1016/j.jacc.2006.08.035. Epub 2006 Nov 28. PMID 17174180
- [Background] Fajadet J, Wijns W, Laarman GJ, Kuck KH, Ormiston J, Munzel T, Popma JJ, Fitzgerald PJ, Bonan R, Kuntz RE; ENDEAVOR II Investigators. Randomized, double-blind, multicenter study of the Endeavor zotarolimus-eluting phosphorylcholine-encapsulated stent for treatment of native coronary artery lesions: clinical and angiographic results of the ENDEAVOR II trial. Circulation. 2006 Aug 22;114(8):798-806. doi: 10.1161/CIRCULATIONAHA.105.591206. Epub 2006 Aug 14. PMID 16908773
- [Derived] Suttorp MJ, Laarman GJ; PRISON III study investigators. A randomized comparison of sirolimus-eluting stent implantation with zotarolimus-eluting stent implantation for the treatment of total coronary occlusions: rationale and design of the PRImary Stenting of Occluded Native coronary arteries III (PRISON III) study. Am Heart J. 2007 Sep;154(3):432-5. doi: 10.1016/j.ahj.2007.04.041. PMID 17719285